CLINICAL TRIAL: NCT00738855
Title: Clinical Impacts of Oral Gastrografin Follow Through in Adhesive Small Bowel Obstruction (SBO).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Amir Fikry, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: oral gastrografin; oral; gastrografin; follow through; in; adhesive SBO.
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-08

CONDITIONS: Small Bowel Obstruction
Keywords: Adhesions; Oral contrast; Exploration
MeSH Terms: conditions — Tissue Adhesions | interventions — Diatrizoate Meglumine; Contrast Media

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Gastrografin group
  Interventions: Other: Oral Gastrografin
- 2 (Placebo Comparator): Control group
  Interventions: Other: Nothing per os

INTERVENTIONS:
Other: Oral Gastrografin — 100 ml of the dye administered through a nasogastric tube
  Other Names: oral contrast
  Arms: 1
Other: Nothing per os — A nasogastric tube
  Other Names: no oral contrast
  Arms: 2

SUMMARY:
Mini abstract :

Altogether 100 patients with 117 episodes of ASBO were randomized into control and gastrografin groups. Eight episodes in eight patients were excluded. Gastrografin group showed a significant decrease of both the time between admission and operation and that of hospital stay .The need for surgery was reduced but statistically insignificant.

DETAILED DESCRIPTION:
Abstract

Background:

Many published studies have shown that Gastrografin can be used for diagnosis post operative acute small bowel obstruction (ASBO) and assessing the need for surgical intervention .However,the studies have reported conflicting results hence the aim of our study to test this hypothesis.

Patients and methods :

Altogether 100 patients with 117 episodes of ASBO were randomized into control and gastrografin groups in a double blinded fashion. Eight episodes in eight patients were excluded due to protocol violation. In Gastrografin group,100 ml of the dye administered through a nasogastric tube and complete obstruction has been considered if the contrast failed to reach the colon on the 24-hour film. Patients were operated on only if they developed signs of strangulation or failed to improve within 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to our surgical department by postoperative SBO were considered for inclusion in this trial.

Exclusion Criteria:

* Age less than 18 years
* Large bowel obstruction
* Recent (within 4 weeks) abdominal surgery
* Ileus
* Cancer peritonitis
* Peritonitis
* Strangulation symptoms and signs
* Obstructed abdominal wall or groin hernia
* Subtotal or total colectomy
* All patients in whom the final diagnosis was not SBO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
resolving | 48 hours

SECONDARY OUTCOMES:
non resolving | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: amir fikry, MD, Principal Investigator — Mansoura University Hospital; ayman mohamed, MD, Study Director — Mansoura University Hospital
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt